CLINICAL TRIAL: NCT05547594
Title: Impact of a Multimodal Prehabilitation Programme on Markers of Health, Quality of Life and the Short and Long Post-surgery Recovery Period in Cancer Patients With Type 2 Diabetes
Brief Title: Prehabilitation in Patients With Cancer and Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Greenwich (Other)
Responsible Party: Principal Investigator, Fernando Naclerio, Professor in Strength Training and Sports Nutrition, University of Greenwich
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UoG_2022_CT2D_Prehab
Record Dates: First submitted 2022-09-12; First posted 2022-09-21 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Cancer; Type 2 Diabetes
Keywords: cancer; Type 2 diabetes; surgery; prehabilitation; recovery; exercise; nutrition; protein; anxiety; quality of life; physical performance
MeSH Terms: conditions — Neoplasms; Diabetes Mellitus, Type 2; Motor Activity; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation (Experimental): Arm undergoing multimodal prehabilitation (physical activity, nutritional education and anxiety management) during the weeks leading up to surgery
  Interventions: Behavioral: Multimodal surgical prehabilitation
- Standard of care (No Intervention): Arm receiving standard of care (no prehabilitation)

INTERVENTIONS:
Behavioral: Multimodal surgical prehabilitation — Participants will be encouraged to engage in regular physical activity (endurance and resistance exercise), eat healthily and undergo cognitive behavioural therapy (the latter only if required) during the weeks prior to surgery.
  Arms: Prehabilitation

SUMMARY:
Surgical prehabilitation refers to pre-operative interventions aimed at increasing patients' physiological reserve so that they can better cope with the stress of surgery, avoid post-operative complications and have a faster recovery after surgery. Multimodal prehabilitation combines different aspects related to a healthy lifestyle including but not limited to; physical activity, nutritional education, anxiety coping strategies, alcohol moderation and smoking cessation. Although these aspects are well known, having a cancer diagnosis and the likelihood of an incoming operation during the weeks after diagnosis, place patients in a situation where they may be more receptive to adopting lifestyle changes aimed at promoting health. Such changes could be incorporated, not just in the short-term in preparation for surgery, but also in the medium- and long-term, improving patients' wellbeing and potentially reducing the risk of cancer reoccurrence and other diseases.

Although the benefits of prehabilitation before surgery are understood, the effects it may have in non-insulin-dependent Type 2 diabetes patients are unknown.

This project aims to: (i) Analyse the effects of a multimodal prehabilitation programme vs. the current National Health Service (NHS) standard approach, on physical performance in cancer patients with non-insulin-dependent Type 2 diabetes prior to surgery. (ii) Explore the impact of the programme on body composition and metabolic markers. (iii) Analyse the programme adherence, markers of well-being and quality of life during a post-surgery period of up to 12 months as well as its effects on clinical outcomes.

DETAILED DESCRIPTION:
This study will take advantage of already existing infrastructures, by approaching a single National Health Service (NHS) hospital in England that is already run a prehabilitation service for its patients. This study will analyse the effect of the prehabilitation programme on a specific group of patients, those with cancer and Type 2 diabetes who do not require insulin as part of their diabetes treatment and who are waiting for surgery.

Surgical prehabilitation refers to interventions done before surgery to increase the patient's overall health and fitness so that they can better cope with the stress of surgery, avoid complications/reduce, and have a faster recovery after surgery. Multimodal prehabilitation combines different aspects related to a healthy lifestyle, including but not limited to; physical activity, nutritional education, anxiety coping strategies, alcohol moderation and smoking cessation.

Multimodal prehabilitation programmes may use a combination of telehealth and face-to-face delivery to provide flexibility according to the preferences of the patients.

The collaboration between the University of Greenwich and NHS will provide an opportunity to measure the impact of the programme on those participants with Type 2 diabetes, beyond variables like weight and fasting blood glucose (i.e., body composition, glycaemic behaviour, blood insulin concentration, immune system markers…).

The hospital prehabilitation team will identify potential study participants (patients with Type 2 diabetes who do not use insulin awaiting surgery) amongst those referred to their service. The prehabilitation team will present the idea of the study to the potential participants and will ask for consent to share their contact details with the sponsor. If consent is received, the researcher will contact them to briefly present to them the possibility of joining the study. This 1st contact will be overseen by the Chief Investigator.

Those who accept to participate in the study will be allocated into 2 different groups. Patients undergoing prehabilitation will join the prehabilitation group of the study, while those declining prehabilitation will join the control group.

Regardless of the group, all patients will undergo the same number of interactions with the researcher:

1. Interview and consent The candidate will be provided with the patient information sheet and explained what they can expect and what will be expected from them if they decide to participate in the study. Candidates will be able to ask questions and, in case they decide to participate, they will sign the participant consent form.
2. Baseline/initial assessment The participant will undergo a number of tests/measurements/questionnaires to obtain information on their physical performance quality of life, body composition, glycaemic markers and immune system markers.

   This assessment will take place a few weeks before surgery before the patient starts prehabilitation (prehab group) or upon joining the study (control group).
3. Assessment before surgery The participant will undergo a number of tests/measurements/questionnaires to obtain information on their physical performance quality of life, body composition, glycaemic markers and immune system markers.

   This assessment will take place a few days before surgery.
4. Assessment 6 weeks after surgery The participant will undergo a number of tests/measurements/questionnaires to obtain information on their physical performance quality of life, body composition, glycaemic markers and immune system markers.

   This assessment will take place 6 weeks after surgery, a time that generally allows the participant to recover enough to be able to move around comfortably and perform some light physical activity
5. Assessment 6 months after surgery The participant will undergo a number of tests/measurements/questionnaires to obtain information on their physical performance quality of life, body composition, glycaemic markers and immune system markers.

   This assessment will take place 6 months after surgery, a time by which the patient will generally be fully recovered, potentially reaching their pre-surgical status, and will have been able to resume their regular day-to-day activity
6. Assessment 12 months after surgery The participant will undergo a number of tests/measurements/questionnaires to obtain information on their physical performance quality of life, body composition, glycaemic markers and immune system markers.

Both groups (prehabilitation and control) will undergo the same previously described assessments. This will allow us to understand and compare how the measured variables change through time in both groups (prehabilitation vs control).

The investigators hypothesise that prehabilitation will improve patients' physical performance prior to surgery and will provide them with a range of tools to help them recover faster and manage their overall health better (including their diabetes control) for at least one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to give consent
* Newly diagnosed with cancer
* Non-insulin-dependent Type 2 diabetes
* Awaiting surgery for cancer

Exclusion Criteria:

* Medical contraindication to engage in physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Short Physical Performance Battery (SPPB) at different time points from baseline to 1 year after surgery | upon enrolment, before surgery, 6 weeks after surgery, 6 and 12 months after surgery
  Group of measures that combines the results of the gait speed, chair stand and balance tests, with scores ranging from 0 (worst performance) to 12 (best performance).

SECONDARY OUTCOMES:
Changes in fasting glucose at different time points from baseline to 1 year after surgery | upon enrolment, before surgery, 6 weeks after surgery, 6 and 12 months after surgery
  Blood fasting glucose obtained via finger prick
Changes in fasting insulin at different time points from baseline to 1 year after surgery | upon enrolment, before surgery, 6 weeks after surgery, 6 and 12 months after surgery
  Blood fasting insulin obtained via finger prick
Changes in BMI at different time points from baseline to 1 year after surgery | upon enrolment, before surgery, 6 weeks after surgery, 6 and 12 months after surgery
  Body mass index
Changes in waist circumference at different time points from baseline to 1 year after surgery | upon enrolment, before surgery, 6 weeks after surgery, 6 and 12 months after surgery
  Waist circumference
Changes in hip circumference at different time points from baseline to 1 year after surgery | upon enrolment, before surgery, 6 weeks after surgery, 6 and 12 months after surgery
  Hip circumferences
Changes in Patient Health Questionnaire-9 (PHQ-9) at different time points from baseline to 1 year after surgery | upon enrolment, before surgery, 6 weeks after surgery, 6 and 12 months after surgery
  Self-administered questionnaires to assess depression severity, with scores ranging from 0 (no depression) to 27 (severe depression)

OTHER OUTCOMES:
Hospital length of stay | 8 weeks after surgery
  Number of days spent in the hospital after surgery
90-day readmission | 90 days after surgery
  Number of readmissions during the 90 days after surgery
Postsurgical complications | 6 months after surgery
  Number of complications after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Naclerio, PhD, Principal Investigator — University of Greenwich
Locations (2):
- United Kingdom (2):
  - School of Human Sciences, University of Greenwich, Avery Hill Campus, Sparrows Farm (Office SF112B), Eltham, England
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wu F, Rotimi O, Laza-Cagigas R, Rampal T. The Feasibility and Effects of a Telehealth-Delivered Home-Based Prehabilitation Program for Cancer Patients during the Pandemic. Curr Oncol. 2021 Jun 17;28(3):2248-2259. doi: 10.3390/curroncol28030207. PMID 34204531